CLINICAL TRIAL: NCT00618839
Title: Open-Label, Controlled, Randomized, Comparative, Dose Escalation Study Of The Safety, Human Immunology, And Efficacy Of StrataGraft™ Skin Tissue (Human Donor Skin) In The Surgical Management Of Complex Skin Defects In Patients Undergoing Sequential Skin Reconstruction Procedures
Brief Title: StrataGraft™ Skin Tissue (Human Donor Skin) In The Surgical Management Of Complex Skin Defects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRATA2001; R44AR047499 (NIH)
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Results first posted 2012-09-10 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2018-12

CONDITIONS: Third Degree Burn; Burns; Wound Infection; Degloving Injury
Keywords: Complex skin defects; Burns; Wound infection; Skin trauma
MeSH Terms: conditions — Burns; Wound Infection; Degloving Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- StrataGraft : cadaver allograft (Experimental): All patients enrolled received StrataGraft skin tissue and an intrapatient control area treated with cadaver allograft in a split-wound design
  Interventions: Biological: StrataGraft Skin Tissue; Procedure: Cadaver allograft

INTERVENTIONS:
Biological: StrataGraft Skin Tissue — StrataGraft™ skin tissue is provided as a suturable circular patch of stratified epithelial tissue composed of a living dermal matrix (containing dermal fibroblasts) overlaid with human epidermal cells (NIKS™ cells).
Procedure: Cadaver allograft — The standard of care for temporary coverage of full thickness skin defects is coverage with cadaver allograft until the wound can be autografted.

SUMMARY:
This pilot Phase I/II clinical study will be conducted at up to three clinical sites.

This is an open-label, randomized, comparative study with a maximum of fifteen (15) patients, each with skin defects. The patients are intended to undergo sequential surgical procedures involving surgical skin debridement and temporary allogeneic (cadaver skin) grafting at various separate or contiguous wound sites. Patients will be randomized within each wound site to one of two test products: cadaver skin or StrataGraft™ skin tissue.

DETAILED DESCRIPTION:
Stratatech has completed a phase I/IIa clinical study to assess the safety and efficacy of escalating amounts of StrataGraft skin tissue in patients with complex skin defects requiring sequential debridement and temporary wound coverage with biological dressing prior to autografting. The specific objectives of this phase I/IIa clinical trial were to assess the safety of StrataGraft skin tissue using a predetermined panel of clinical and laboratory endpoints and assess the efficacy of StrataGraft skin tissue by comparing the ability of StrataGraft skin tissue to the standard of care, human cadaver skin, to condition complex skin defects for subsequent autografting. In three cohorts of five patients each, the maximum amount of StrataGraft skin tissue applied to excised full-thickness skin wounds was increased sequentially from 0.5% to 1.0%, and then to 1.5% TBSA. Equivalent study wound areas on each subject were treated with StrataGraft or cadaver allograft for one week, at which time the allograft tissues were removed and the wound bed was evaluated. Infection and appearance of the temporary allogeneic skin tissue were evaluated at every study session until autograft placement. The wound was covered with split-thickness skin autografts when the wound was judged ready to accept an autograft. Autograft take was assessed two weeks after autograft placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged greater than 18 yrs.
* Patients with complex skin defects requiring sequential debridement under anesthesia with temporary biological dressing (allogeneic grafting) prior to autografting
* Full-thickness skin defects
* Informed consent

Exclusion Criteria:

* Prisoners
* Pregnant (positive urinary pregnancy in women of child-bearing potential at Visit#1) or lactating females
* Immunosuppressive therapy
* Infection with Human Immunodeficiency Virus
* Venous stasis ulcers of the lower leg
* Diabetic foot ulcers
* Donor site wounds
* Wounds of less than 5% body surface area
* Wounds of the hands, face, and feet (although such wound surface areas can be counted toward total injured BSA)
* Prior entry into this study
* Expected survival of less than 3 months
* Concomitant processes sustained contemporaneously with the dermal injury (e.g., inhalational injury requiring ventilation, electrical injury with cardiac damage or arrhythmia, sepsis, other serious or unstabilized organ damage from trauma, etc.)
* Use of an investigational agent within 30 days
* Active malignancy
* Clinical evidence of malnutrition
* Clinically significant renal, hepatic, cardiac, pulmonary, or neurological impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Stratatech, Inc., a Mallinckrodt Pharmaceeuticals
Locations (2):
- United States (2):
  - Arizona Burn & Trauma Center, Phoenix, Arizona
  - University of Wisconsin-Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Result] Schurr MJ, Foster KN, Centanni JM, Comer AR, Wicks A, Gibson AL, Thomas-Virnig CL, Schlosser SJ, Faucher LD, Lokuta MA, Allen-Hoffmann BL. Phase I/II clinical evaluation of StrataGraft: a consistent, pathogen-free human skin substitute. J Trauma. 2009 Mar;66(3):866-73; discussion 873-4. doi: 10.1097/TA.0b013e31819849d6. PMID 19276766
- [Result] Centanni JM, Straseski JA, Wicks A, Hank JA, Rasmussen CA, Lokuta MA, Schurr MJ, Foster KN, Faucher LD, Caruso DM, Comer AR, Allen-Hoffmann BL. StrataGraft skin substitute is well-tolerated and is not acutely immunogenic in patients with traumatic wounds: results from a prospective, randomized, controlled dose escalation trial. Ann Surg. 2011 Apr;253(4):672-83. doi: 10.1097/SLA.0b013e318210f3bd. PMID 21475006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study evaluated autograft take and infection in 15 patients with full-thickness skin defects who required sequential surgical procedures. Subjects had surgical excision and temporary placement of StrataGraft and cadaver allograft. The trial was conducted at the University of Wisconsin Hospital and the Arizona Burn Center.
Pre-assignment Details: All subjects were treated with both StrataGraft and cadaver allograft in a split-wound design. The half-wound sites were randomized to receive StrataGraft or cadaver allograft.
Groups:
- StrataGraft : Cadaver Allograft: Wounds were excised and the half-wound sites were randomized to receive StrataGraft skin tissue or cadaver allograft for 7 days until the wounds were ready for autografting.
Period: Overall Study
Arm/Group | StrataGraft : Cadaver Allograft
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | StrataGraft : Cadaver Allograft
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Autograft Take on Wounds Prepared by StrataGraft™ Skin Tissue.
Description: The percentage take of the autografted area on each treatment site based on clinical judgement of visual and tactile assessments two weeks after autografting of wounds that had been temporarily covered with StrataGraft skin tissue.
Time Frame: two weeks post-autografting
Population: Intrapatient treatment sites were randomized such that each half of the wound site received StrataGraft and the other half received cadaver skin. Therefore, each patient received StrataGraft and cadaver allograft.
Measure: Mean (Standard Deviation); unit: Percent Area of Autograft Take (%)
Groups:
- StrataGraft Skin Tissue: StrataGraft skin tissue is a fully-differentiated tissue which exhibits barrier function comparable to that of intact human skin. StrataGraft consists of an epidermal layer of fully-stratified human keratinocytes growing on a dermal layer which is comprised of human fibroblasts embedded in a collagen matrix. StrataGraft skin tissue is a tough, suturable, meshable tissue product that is manufactured with a surface area of 44 cm2. StrataGraft tissue is not intended to be a patient-specific product but rather to provide an allogeneic skin substitute which reproduces many of the structural and biological properties of normal human skin and is anticipated to serve as a biological wound dressing.
- Cadaver Skin: The current standard of care for the management of severe burns or other major skin trauma is temporary coverage of the wound with cadaver skin followed by autografting once once sufficient donor skin is available for autografting. Excised wounds are covered temporarily with cadaver skin to reduce fluid loss and infection. In addition to preventing excessive dehydration, restoration of a permeability barrier maintains a moist wound environment which promotes wound healing. However, there is inconsistent availability of freshly-harvested cadaver grafts. In addition, the quality of cadaver skin is variable- cadaver skin is often contaminated and if cadaver skin had undergone prolonged storage or freezing this reduces the viability of cadaver skin.
Arm/Group | StrataGraft Skin Tissue | Cadaver Skin
Number analyzed (Participants) | 15 | 15
Percent Area of Autograft Take (%) | 97.7 (6.78) | 96.7 (10.47)

2. Secondary Outcome: Appearance of Allograft Tissues
Description: The following three point scale was used to assess the condition of skin allografts: pink and adherent (2 points); either pink or adherent but not both (1 point); or neither pink nor adherent (0 points).
Time Frame: StrataGraft and cadaver allograft appearance were performed every other day after placement and at the time of allograft removal and the values averaged for each subject.
Population: Treatment for each patient was randomized such that each half of the wound site received StrataGraft or cadaver skin. Therefore, each patient received StrataGraft and cadaver allograft.
Measure: Mean (Standard Error); unit: points
Groups:
- StrataGraft: StrataGraft skin tissue is a fully-differentiated tissue which exhibits barrier function comparable to that of intact human skin. StrataGraft consists of an epidermal layer of fully-stratified human keratinocytes growing on a dermal layer which is comprised of human fibroblasts embedded in a collagen matrix. StrataGraft skin tissue is a tough, suturable, meshable tissue product that is manufactured with a surface area of 44 cm2. StrataGraft tissue is not intended to be a patient-specific product but rather to provide an allogeneic skin substitute which reproduces many of the structural and biological properties of normal human skin and is anticipated to serve as a biological wound dressing.
- Cadaver Skin: The current standard of care for the management of severe burns or other major skin trauma is temporary coverage of the wound with cadaver skin followed by subsequent autografting once the wound bed has become healthy enough to accept an autograft. Excised wounds are covered temporarily with cadaver skin to reduce fluid loss and infection. In addition to preventing excessive dehydration, restoration of a permeability barrier maintains a moist wound environment which promotes wound healing. However, there is inconsistent availability of freshly-harvested cadaver grafts. In addition, the quality of cadaver skin is variable- cadaver skin is often contaminated and if cadaver skin had undergone prolonged storage or freezing this reduces the viability of cadaver skin.
Arm/Group | StrataGraft | Cadaver Skin
Number analyzed (Participants) | 15 | 15
points | 1.70 (0.62) | 1.49 (0.65)

3. Secondary Outcome: Viability of Allograft Tissues
Description: Immunohistochemical staining for Ki67, a protein expressed only in proliferating cells.
Time Frame: At the time of allograft removal (~7 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: Ki67 positive cells/ total cells
Arm/Group | StrataGraft | Cadaver Skin
Number analyzed (Participants) | 15 | 15
Ki67 positive cells/ total cells | 0.567 (0.175) [0.283 to 0.807] | 0.189 (0.315) [0.015 to 0.959]

ADVERSE EVENTS:
Arm/Group | StrataGraft : Cadaver Allograft
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StrataGraft : Cadaver Allograft (N=15)
IMPAIRED HEALING (General disorders) | 1 (1) — Poor graft healing found approximately 48 days following autograft placement. This event was judged to be unrelated to treatment with StrataGraft skin tissue.
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) — The bilateral pulmonary embolism was judged unrelated to treatment with StrataGraft skin tissue.
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) — The right knee effusion was judged unrelated to treatment with StrataGraft skin tissue.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StrataGraft : Cadaver Allograft (N=15)
INFECTION (Infections and infestations) | 9 (13) — There was no difference in infection between StrataGraft and cadaver skin. 1 subject was visually infected at both sites and 2 subjects had laboratory evidence of infection at both sites. Infection was judged unrelated to StrataGraft skin tissue.
CONSTIPATION (Gastrointestinal disorders) | 8 (10) — All adverse events (AE) were judged unrelated to treatment with StrataGraft skin tissue.
NAUSEA (Gastrointestinal disorders) | 8 (9) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ANXIETY (Psychiatric disorders) | 6 (8) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DIARRHOEA (Gastrointestinal disorders) | 7 (8) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
INSOMNIA (Psychiatric disorders) | 8 (8) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
AGITATION (Psychiatric disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ALBUMIN GLOBULIN RATIO DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
APHONIA (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ASPARTATE AMINOTRANSFERASE DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ASTHENIA (General disorders) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLISTER (Skin and subcutaneous tissue disorders) | 2 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD ALBUMIN DECREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD BILIRUBIN DECREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD CARBON DIOXIDE DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD CHLORIDE DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD CHLORIDE INCREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD CREATININE DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD CULTURE POSITIVE (Investigations) | 3 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD MAGNESIUM INCREASED (Investigations) | 4 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD PHOSPHOROUS ELEVATED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD PHOSPHORUS INCREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD POTASSIUM INCREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD UREA DECREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BLOOD UREA INCREASED (Investigations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 2 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
BURNING SENSATION (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
CELLULITIS (Infections and infestations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
CHILLS (General disorders) | 2 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
CONFUSIONAL STATE (Psychiatric disorders) | 3 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
CULTURE POSITIVE (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
CYST (General disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DEPRESSION (Psychiatric disorders) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DIZZINESS (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
DYSURIA (Renal and urinary disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ECTROPION (Eye disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ELEVATED PHOSPHOROUS (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ESCHAR (Injury, poisoning and procedural complications) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
EXTRASKELETAL OSSIFICATION (Musculoskeletal and connective tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
EYE IRRITATION (Eye disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
FLATULENCE (Gastrointestinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
GLOBULINS INCREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HAEMATOCRIT DECREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HAEMOGLOBIN DECREASED (Investigations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HERPES SIMPLEX (Infections and infestations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HIGH DENSITY LIPOPROTEIN DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPERAESTHESIA (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPERTENSION (Vascular disorders) | 4 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPERTROPHIC SCAR (Skin and subcutaneous tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOAESTHESIA (Nervous system disorders) | 2 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 5 (5) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (5) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOTENSION (Vascular disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
HYPOTHERMIA (General disorders) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
IMPAIRED HEALING (General disorders) | 1 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
LIVEDO RETICULARIS (Skin and subcutaneous tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
MALNUTRITION (Metabolism and nutrition disorders) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
MEAN PLATELET VOLUME DECREASED (Investigations) | 4 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
MICROSTOMIA (Congenital, familial and genetic disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
MONOCYTE COUNT INCREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
NEURALGIA (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
NEUTROPHIL COUNT INCREASED (Investigations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
NOCTURIA (Renal and urinary disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
OEDEMA (General disorders) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
OEDEMA PERIPHERAL (General disorders) | 2 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
OPEN WOUND (Injury, poisoning and procedural complications) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PARAESTHESIA (Nervous system disorders) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PCO2 DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PERONEAL NERVE PALSY (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PLATELET COUNT INCREASED (Investigations) | 8 (8) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PLATELET MORPHOLOGY ABNORMAL (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PNEUMONIA (Infections and infestations) | 5 (5) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 1 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PROTHROMBIN TIME PROLONGED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (5) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PRURITUS ANI (Gastrointestinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PURULENT DISCHARGE (Infections and infestations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
PYREXIA (General disorders) | 3 (5) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RADIAL NERVE PALSY (Nervous system disorders) | 1 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RASH (Skin and subcutaneous tissue disorders) | 4 (4) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RED BLOOD CELL COUNT DECREASED (Investigations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RED BLOOD CELLS URINE (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RED CELL DISTRIBUTION WIDTH INCREASED (Investigations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
RESTLESSNESS (Psychiatric disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
SEPTIC SHOCK (Infections and infestations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
SINUSITIS (Infections and infestations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
SOMNOLENCE (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
TACHYCARDIA (Cardiac disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
TENDERNESS (General disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
TOOTH DISORDER (Gastrointestinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
TRANSFERRIN DECREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
TREMOR (Nervous system disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
ULCER (Skin and subcutaneous tissue disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
URINARY RETENTION (Renal and urinary disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
URINE OUTPUT DECREASED (Investigations) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
VOMITING (Gastrointestinal disorders) | 3 (6) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 3 (3) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
WOUND (Injury, poisoning and procedural complications) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
WOUND CLOSURE (Surgical and medical procedures) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.
WOUND INFECTION (Infections and infestations) | 2 (2) — All AE were judged to be unrelated to treatment with StrataGraft skin tissue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No